CLINICAL TRIAL: NCT05253300
Title: Laparoskopik Kolesistektomi Ameliyatı Sonrası Omuz Ağrısının Giderilmesinde Semi Rekümbent Pozisyonunun Etkisi
Brief Title: Effect of Semi-recumbent Position on Treatment of Shoulder Pain Seen After Laparoscopic Cholecystectomy
Acronym: SRPSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Yilmaz Sahin (Other)
Responsible Party: Sponsor-Investigator, Sibel Yilmaz Sahin, Assistant professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SRPShoulderPain
Record Dates: First submitted 2022-01-12; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Shoulder Pain
Keywords: laparoscopic cholecystectomy; shoulder pain; semi-recumbent position; pain
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Intervention Model Description: The type of this study is a quasi-experimental clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi Recumbent (Experimental): The patients' vital signs, pain and analgesic drug use were recorded in the "Pain Follow-up Form" at the time they came to the clinic, at the 6th and 12th hours after the surgery, by recording from the end-of-operation file. In case the patient had pain, the time when the pain started was recorded, the experimental group was given the semi-recumbent position with analgesic drug and the patient was asked to maintain this position for 2 hours. If the patient has pain again, this position is given again. "Patient Satisfaction Evaluation Form" was filled in at the 12th hour after the surgery for the patients in the experimental group.
  Interventions: Other: Positioning the patient
- Control (No Intervention): The patients' vital signs, pain and analgesic drug use were recorded in the "Pain Follow-up Form" at the time they came to the clinic, at the 6th and 12th hours after the surgery, by recording from the end-of-operation file. In case the patient has pain, the time when the patients' pain started was recorded, and only analgesic medication was administered to the control group.

INTERVENTIONS:
Other: Positioning the patient — The patients' vital signs, pain and analgesic drug use were recorded in the "Pain Follow-up Form" at the time they came to the clinic, at the 6th and 12th hours after the surgery, by recording from the end-of-operation file. In case the patient had pain, the time when the pain started was recorded, the experimental group was given the semi-recumbent position with analgesic drug and the patient was asked to maintain this position for 2 hours. If the patient has pain again, this position is given again. "Patient Satisfaction Evaluation Form" was filled in at the 12th hour after the surgery for the patients in the experimental group.
  Arms: Semi Recumbent

SUMMARY:
This study was carried out to determine the effect of placing the semi-recumbent position in reducing pain in patients who developed shoulder pain after laparoscopic cholecystectomy.

HO: The application of the semi-recumbent position to patients who develop shoulder pain after laparoscopic cholecystectomy has no effect on reducing pain.

H1: The application of semi-recumbent position in patients who develop shoulder pain after laparoscopic cholecystectomy has an effect on reducing pain.

DETAILED DESCRIPTION:
In addition to pharmacological interventions for the relief of postoperative complications such as pain in patients undergoing laparoscopic cholecystectomy, non-pharmacological applications; It is evaluated that it will be beneficial in increasing patient satisfaction, reducing the need for analgesic drugs, reducing the cost of hospitalization due to the side effects of drugs and increasing the quality of care. With the results of this research, it is evaluated that the effect of positioning, which is one of the independent activities of nurses who base their care on evidence-based practices, on pain will be beneficial to increase the evidence-based nursing knowledge in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Those who had surgery with laparoscopic cholecystectomy
* Those between the ages of 18-65,
* Patients in ASA I-II group
* Patients undergoing general anesthesia

Exclusion Criteria:

* Epidural analgesia after surgery
* Patients with reactive airway diseases such as chronic obstructive pulmonary disease (COPD), Bronchitis, Emphysema
* Conversion to open abdominal surgery during laparoscopic cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-07-24 (Actual)

PRIMARY OUTCOMES:
Pain Severity | arrival time at the clinic (approximately the first two hours postoperatively)
  Pain evaluated with numerical rating scale (NRS). A numerical rating scale requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Pain Region | arrival time at the clinic (approximately the first two hours postoperatively)
  Description of pain region as
  1. Right shoulder
  2. Left shoulder
  3. Both shoulder
  4. Back
  5. Incision
  6. Other
Pain Severity | postoperative 6th hour
  Pain evaluated with numerical rating scale (NRS). A numerical rating scale requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Pain Region | postoperative 6th hour
  Description of pain region as
  1. Right shoulder
  2. Left shoulder
  3. Both shoulder
  4. Back
  5. Incision
  6. Other
Pain Severity | postoperative 12th hour
  Pain evaluated with numerical rating scale (NRS). A numerical rating scale requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Pain Region | postoperative 12th hour
  Description of pain region as
  1. Right shoulder
  2. Left shoulder
  3. Both shoulder
  4. Back
  5. Incision
  6. Other

SECONDARY OUTCOMES:
Use Analgesia | postoperatarrival time at the clinic (approximately the first two hours postoperatively)
  Number of Analgesia used to reduce pain since arrival
Use Analgesia | postoperative 6th hour
  Number of Analgesia used to reduce pain between arrival time and 6th hour
Use Analgesia | postoperative 12th hour
  Number of Analgesia used to reduce pain between 6th hour and 12th hour

OTHER OUTCOMES:
patient's satisfaction with the given position | postoperative 12th hour
  Used Yes or No question to evaluate if patient were satisfied with the semi-recumbent position to prevent post-operative shoulder pain and Whether they think the semi-recumbent position is beneficial.
  Numerical rating scale (NRS) were used to evaluate how satisfied they are with the semi-recumbent position to avoid surgery-related shoulder pain and How much discomfort they felt during their stay in the semi-recumbent position. NRS of 0 to10 were used and rated as 0 is not at all and 10 is very much

CONTACTS AND LOCATIONS:
Overall Officials: Sibel YILMAZ SAHIN, Asst. Prof., Study Chair — Gulhane Faculty of Nursing, University of Health Sciences, Ankara, Turkey
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749
- [Background] Pasquier EK, Andersson E. Pulmonary recruitment maneuver reduces pain after laparoscopic bariatric surgery: a randomized controlled clinical trial. Surg Obes Relat Dis. 2018 Mar;14(3):386-392. doi: 10.1016/j.soard.2017.11.017. Epub 2017 Nov 22. PMID 29290563
- [Background] Aydemir O, Aslan FE, Karabacak U, Akdas O. The Effect of Exaggerated Lithotomy Position on Shoulder Pain after Laparoscopic Cholecystectomy. Pain Manag Nurs. 2018 Dec;19(6):663-670. doi: 10.1016/j.pmn.2018.04.012. Epub 2018 Jun 19. PMID 29934129